CLINICAL TRIAL: NCT03633539
Title: Multi-center Prospective Randomized Controlled Study of the Single-incision Laparoscopic Surgery Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Brief Title: Single-incision Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Acronym: mSILSC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No research funds were raised
Sponsor: Ruijin Hospital (Other)
Collaborators: Changhai Hospital (Other); Fudan University (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-mSILSC-2018
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Colonic Neoplasms; Rectal Neoplasms; Colon Disease; Colon Cancer; Rectal Cancer; Rectal Diseases
Keywords: SILS; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Colonic Diseases; Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Laparoscopic Surgery (Active Comparator): Patients with colorectal cancer undergo conventional laparoscopic surgery（multi-ports）.
  Interventions: Procedure: Conventional Laparoscopic Surgery
- Single-incision Laparoscopic Surgery (Experimental): Patients with colorectal cancer undergo single-incision laparoscopic surgery.
  Interventions: Procedure: Single-incision Laparoscopic Surgery

INTERVENTIONS:
Procedure: Single-incision Laparoscopic Surgery — Patients undergo single-incision laparoscopic surgery. In this group，the surgery is performed through a transumbilical port. The surgeon will adjust surgical position to expose the operative field with the help of gravity. Besides，hand over hand cross and parallel techniques are needed to achieve the SILS. All the other operative procedures are the same as conventional laparoscopic surgery.
  Other Names: SILSC
  Arms: Single-incision Laparoscopic Surgery
Procedure: Conventional Laparoscopic Surgery — Patients undergo conventional laparoscopic surgery. In this group，the surgery is performed through 3-5 ports according to the surgeons habits and specific conditions.
  Other Names: CLSC
  Arms: Conventional Laparoscopic Surgery

SUMMARY:
This study is designed to evaluate the short-term and long-term results after single incision laparoscopic surgery for colorectal cancer（SILSC） compared with conventional laparoscopic surgery for colorectal cancer（CLSC）.

DETAILED DESCRIPTION:
In order to improve cosmetic effect and reduce postoperative pain, single-incision laparoscopic surgery (SILS) is attracting increasing attention. SILS is considered to be the next major advance in the progress of minimally invasive surgical approaches to colorectal disease that is more feasible in generalized use. In most previous studies, SILS for colorectal cancer was feasible and short-term safe compared to conventional laparoscopic surgery (CLS) . However, there is still controversy over its potential better cosmetic effect and less postoperative pain. Moreover, the long-term oncologic outcomes are still inconclusive as only a few studies showed long-term survival data. Up to now, most studies were limited to their retrospective nature and small samples. So more studies, especially large-scale, randomized controlled trials are needed to establish the best indications for SILS for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* 18 years < age ≤85 years
* Tumor located in colon and high rectum ( the lower border of the tumor is above the peritoneal reflection)
* Pathological colorectal carcinoma
* Clinically diagnosed cT1-4aN0-2 M0 lesions according to the 8th Edition of AJCC Cancer Staging Manual
* Tumor size of 5 cm or less
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >35 kg/m2
* The lower border of the tumor is located distal to the peritoneal reflection
* Pregnant woman or lactating woman
* Severe mental disease
* Previous abdominal surgery（except appendectomy and cholecystotomy）
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after surgery
  Postoperative complications rate 30 days after surgery

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Incision length | intraoperative
  Incision length（centimeters，cm）
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Incisal margin | 14 days after surgery
  Length of proximal and distal margin （centimeters，cm）
Tumor size | 14 days after surgery
  The diameter of tumors（centimeters，cm）
Length of stay | 1-14 days after surgery
  Duration of hospital stay（days after surgery）
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and soft diet （hours after surgery）
Pain score | 1-3 days after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3 and the day of discharge
3-year disease free survival rate | 36 months after surgery
  3-year disease free survival rate
5-year overall survival rate | 60 months after surgery
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Kun Liu, MD, Study Chair — Ruijin Hospitla North
Locations (1):
- Ruijin Hospital North, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Song Z, Li Y, Liu K, Jiang Y, Shi Y, Ji X, Zhang T, Wu H, Shi Y, Zhao R. Clinical and oncologic outcomes of single-incision laparoscopic surgery for right colon cancer: a propensity score matching analysis. Surg Endosc. 2019 Apr;33(4):1117-1123. doi: 10.1007/s00464-018-6370-2. Epub 2018 Jul 24. PMID 30043168